CLINICAL TRIAL: NCT02487914
Title: Iontophoresis Effects on Senses
Brief Title: Evaluation of Pressure Sense Threshold and Tactile Sensation After Lidocaine Iontophoresis Using Interferential Current
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Motealleh, Dr. Amin Kordi Yoosefinejad, Shiraz University of Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 386
Record Dates: First submitted 2015-06-15; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Interferential Current Drug Delivery
Keywords: Drug Delivery; Iontophoresis; Lidocaine; Pressure; Tactile perception
MeSH Terms: interventions — Lidocaine; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- lidocaine iontophoresis using interferential current (Active Comparator): the threshold of pressure, tactile,and pain thresholds were evaluated after the iontophoresis of Lidocaine using interferential current.
  Interventions: Device: iontophoresis of Lidocaine 10% with interferential current (Dynatron 438)
- interferential current (Active Comparator): the threshold of pressure, tactile,and pain thresholds were evaluated after the application of interferential current.
  Interventions: Device: interferential current
- lidocaine (Active Comparator): the threshold of pressure, tactile,and pain thresholds were evaluated after the application of topical Lidocaine.
  Interventions: Drug: Lidocaine 10% was sprayed at the identified region

INTERVENTIONS:
Device: iontophoresis of Lidocaine 10% with interferential current (Dynatron 438) — drug delivery through interferential current.
  Other Names: Dynatron 438, Enraf Nonius Comp., Netherlands
  Arms: lidocaine iontophoresis using interferential current
Drug: Lidocaine 10% was sprayed at the identified region
  Other Names: Xylocaine 10% spray, AstraZeneca, Korea
  Arms: lidocaine
Device: interferential current
  Other Names: Dynatron 438, Enraf Nonius Comp., Netherlands
  Arms: interferential current

SUMMARY:
Drug delivery is conducted through various methods such as injection, phonophoresis, and iontophoresis. Iontophoresis is defined as the noninvasive delivery of active ions through epidermis using direct current. The direct current has some disadvantages such as skin burning and limited time of application. Interferential current is a kind of alternating currents without limitations of direct current; so the purpose of this study was to investigate and compare the effects of Lidocaine, interferential current and Lidocaine iontophoresis using interferential current.

DETAILED DESCRIPTION:
Pressure, tactile, and pain thresholds were evaluated before and after the application of Lidocaine, interferential current and Lidocaine iontophoresis using interferential current. Pressure threshold was investigated with a Pesula. Pesula is a pen-like scaled mechanical device that measures the skin pressure threshold. Pesula was pressed to the skin and pressure threshold was measured in mm. Pain and tactile thresholds were investigated using an electrical stimulator.The intensity was gradually increased to the extent that the participant reported a tingling sensation. The displayed intensity was considered as the tactile sense threshold. Then, the intensity was increased to the extent to be intolerable for the participant and this intensity was considered as the maximum pain threshold. The thresholds were recorded in milliampere.

Lidocaine iontophoresis using interferential current can increase perception threshold of pain, and pressure sense more significantly in comparison to the application of Lidocaine and interferential current alone.

ELIGIBILITY:
Inclusion Criteria:

* healthy women with age between 18 and 25 years old

Exclusion Criteria:

* Systemic disorders,
* neuro-muscular diseases such as diabetes and all forms of neuropathies,
* and use of narcoleptic drugs which may contaminate the results.
* Also, none of the participants were on their menstrual cycle.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
pain threshold- evaluated by increasing intensity of interferential current. | up to one week
  pain threshold to increasing intensity of interferential current.

SECONDARY OUTCOMES:
tactile threshold- evaluated by exact perception of the lowest level of interferential current | up to one week
  exact perception of the lowest level of interferential current
pressure threshold- evaluated by Pesula | up to one week
  Pesula was used to evaluate tactile threshold.

CONTACTS AND LOCATIONS:
Overall Officials: alireza motealleh, PhD, PT, Study Director — Shiraz University of Medical Sciences
Locations (1):
- School of Rehabilitation, Shiraz, Fars, Iran

REFERENCES:
- [Background] Baskurt F, Ozcan A, Algun C. Comparison of effects of phonophoresis and iontophoresis of naproxen in the treatment of lateral epicondylitis. Clin Rehabil. 2003 Feb;17(1):96-100. doi: 10.1191/0269215503cr588oa. PMID 12617384
- [Background] Ebrahimi S, Abbasnia K, Motealleh A, Kooroshfard N, Kamali F, Ghaffarinezhad F. Effect of lidocaine phonophoresis on sensory blockade: pulsed or continuous mode of therapeutic ultrasound? Physiotherapy. 2012 Mar;98(1):57-63. doi: 10.1016/j.physio.2011.01.009. PMID 22265386
- [Background] Gokoglu F, Findikoglu G, Yorgancoglu ZR, Okumus M, Ceceli E, Kocaoglu S. Evaluation of iontophoresis and local corticosteroid injection in the treatment of carpal tunnel syndrome. Am J Phys Med Rehabil. 2005 Feb;84(2):92-6. doi: 10.1097/01.phm.0000151942.49031.dd. PMID 15668556
- [Background] Pal B, Morris J. Perceived risks of joint infection following intra-articular corticosteroid injections: a survey of rheumatologists. Clin Rheumatol. 1999;18(3):264-5. doi: 10.1007/s100670050098. PMID 11206357
- [Background] Jadoul A, Bouwstra J, Preat V V. Effects of iontophoresis and electroporation on the stratum corneum. Review of the biophysical studies. Adv Drug Deliv Rev. 1999 Jan 4;35(1):89-105. doi: 10.1016/s0169-409x(98)00065-9. PMID 10837691
- [Background] Jadoul A, Doucet J, Durand D, Preat V. Modifications induced on stratum corneum structure after in vitro iontophoresis; ATR-FTIR and X-ray scattering studies. J. Controlled Release 42: 165-173,1996.
- [Background] Thysman S, Van Neste D, Preat V. Noninvasive investigation of human skin after in vivo iontophoresis. Skin Pharmacol. 1995;8(5):229-36. doi: 10.1159/000211352. PMID 8527154
- [Background] Costello CT, Jeske AH. Iontophoresis: applications in transdermal medication delivery. Phys Ther. 1995 Jun;75(6):554-63. doi: 10.1093/ptj/75.6.554. PMID 7770500
- [Background] Singh P, Maibach HI. Iontophoresis in drug delivery: basic principles and applications. Crit Rev Ther Drug Carrier Syst. 1994;11(2-3):161-213. PMID 7600587
- [Background] Panzade P, Puranik P. Iontophoresis: A Functional Approach for Enhancement of Transdermal Drug Delivery. Asian Journal of Biomedical and Pharmaceutical Sciences 2(11): 1-8, 2012.
- [Background] Banga AK, Chien YW. Hydrogel-based iontotherapeutic delivery devices for transdermal delivery of peptide/protein drugs. Pharm Res. 1993 May;10(5):697-702. doi: 10.1023/a:1018955631835. PMID 8321834
- [Background] Gupta SK, Bernstein KJ, Noorduin H, Van Peer A, Sathyan G, Haak R. Fentanyl delivery from an electrotransport system: delivery is a function of total current, not duration of current. J Clin Pharmacol. 1998 Oct;38(10):951-8. doi: 10.1002/j.1552-4604.1998.tb04392.x. PMID 9807977
- [Background] Lvovich VF, Matthews E, Riga AT, Kaza L. AC electrokinetic platform for iontophoretic transdermal drug delivery. J Control Release. 2010 Jul 14;145(2):134-40. doi: 10.1016/j.jconrel.2010.04.015. Epub 2010 Apr 24. PMID 20420867
- [Background] Reinauer S, Neusser A, Schauf G, Holzle E. Iontophoresis with alternating current and direct current offset (AC/DC iontophoresis): a new approach for the treatment of hyperhidrosis. Br J Dermatol. 1993 Aug;129(2):166-9. doi: 10.1111/j.1365-2133.1993.tb03521.x. PMID 7654577
- [Background] Ganne JM. Interferential therapy. Aust J Physiother. 1976 Sep;22(3):101-10. doi: 10.1016/S0004-9514(14)61005-9. PMID 25026222
- [Background] Jorge S, Parada CA, Ferreira SH, Tambeli CH. Interferential therapy produces antinociception during application in various models of inflammatory pain. Phys Ther. 2006 Jun;86(6):800-8. PMID 16737405
- [Background] Watson T. The role of electrotherapy in contemporary physiotherapy practice. Man Ther. 2000 Aug;5(3):132-41. doi: 10.1054/math.2000.0363. PMID 11034883
- [Background] Bhatia G, Banga AK. Effect of modulated alternating and direct current iontophoresis on transdermal delivery of lidocaine hydrochloride. Biomed Res Int. 2014;2014:537941. doi: 10.1155/2014/537941. Epub 2014 May 15. PMID 24959580
- [Background] Hayashi S, Ogami S, Shibaji T, Umino M. Lidocaine transport through a cellophane membrane by alternating current iontophoresis with a duty cycle. Bioelectrochemistry. 2009 Feb;74(2):315-22. doi: 10.1016/j.bioelechem.2008.11.007. Epub 2008 Nov 30. PMID 19110474
- [Background] Yan G, Xu Q, Anissimov YG, Hao J, Higuchi WI, Li SK. Alternating current (AC) iontophoretic transport across human epidermal membrane: effects of AC frequency and amplitude. Pharm Res. 2008 Mar;25(3):616-24. doi: 10.1007/s11095-007-9405-2. Epub 2007 Aug 17. PMID 17703345
- [Background] Yamazaki Y, Umino M, Fukayama H, Shimada M. The effect of alternating current iontophoresis on rats with the chronic constriction injury to the infraorbital nerve. Int J Dent. 2012;2012:405292. doi: 10.1155/2012/405292. Epub 2012 May 23. PMID 22675357
- [Background] Kandell ER, Schwartz JH, Jessell TM. Principles of neural science 2000. 4th edition.
- [Result] Viscusi ER, Witkowski TA. Iontophoresis: the process behind noninvasive drug delivery. Reg Anesth Pain Med. 2005 May-Jun;30(3):292-4. doi: 10.1016/j.rapm.2004.12.002. No abstract available. PMID 15898033